CLINICAL TRIAL: NCT01719211
Title: Genetic Basis of Mitral Valve Prolapse
Acronym: MVP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Leducq Foundation (Other)
Responsible Party: Principal Investigator, Robert A. Levine, MD, Cardiologist, Massachusetts General Hospital
Other Study IDs: 1999-p-007948
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Mitral Valve Prolapse
Keywords: MVP, mitral valve
MeSH Terms: conditions — Mitral Valve Prolapse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators have successfully identified two novel genetic loci for MVP on chromosomes 11 and 13 and are searching for altered genes in these regions. This requires recruiting large families who may have MVP linked to these or other chromosomes; and obtaining DNA samples from 1,000-1,500 individually affected patients to study the relation between DNA markers throughout the genome and MVP. It is our expectation that the results of this study will lead to the discovery of gene(s) responsible for MVP. This will lead to improved understanding of the disease and, in turn, improved ability to treat and prevent progression in genetically susceptible individuals.

DETAILED DESCRIPTION:
This is a genome-wide association study.

ELIGIBILITY:
Inclusion Criteria:

* Mitral valve prolapse

Exclusion Criteria:

* Other mitral valve diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for 2D echo for MVP
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 1999-01; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Discovery of the genetic basis of Mitral Valve Prolapse | 5 years
  Genome-wide association

CONTACTS AND LOCATIONS:
Overall Officials: robert a levine, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mass General Hospital, Boston, Massachusetts, United States